CLINICAL TRIAL: NCT04854785
Title: Imaging Neuroinflammation in COVID-19 and Persistent Depression With/Without Other Neuropsychiatric Symptoms
Brief Title: Neuroinflammation in COVID-19 and Depression
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Other Study IDs: 177/2020
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Episode; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — brain scan; also saliva, whole blood, plasma and serum samples will be kept for analysis of genotype, peripheral inflammatory markers and protein binding in relation to brain scan
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (3):
- DNP-mild: Participants that have recovered from mild COVID-19 respiratory symptoms and have a new onset major depressive episode (MDE).
  Interventions: Other: [18F]FEPPA PET scan; Other: [11C]SL25.1188 PET scan
- DNP-moderate: Participants that have recovered from moderate COVID-19 respiratory symptoms and have a new onset major depressive episode (MDE).
  Interventions: Other: [18F]FEPPA PET scan; Other: [11C]SL25.1188 PET scan
- Healthy Control Participants: Participants in good physical health, age- and sex-matched to Group 1 and 2 participants.
  Interventions: Other: [18F]FEPPA PET scan; Other: [11C]SL25.1188 PET scan

INTERVENTIONS:
Other: [18F]FEPPA PET scan — One [18F]FEPPA PET for TSPO VT, and one MRI scan
Other: [11C]SL25.1188 PET scan — One [11C]SL25.1188 PET scan for MAO-B VT, and one MRI scan

SUMMARY:
The purpose of this study is to use state of the art brain imaging technology to investigate neuroinflammation in participants with depression after the respiratory symptoms of coronavirus disease 2019 (COVID-19) have passed.

DETAILED DESCRIPTION:
Participants will undergo two positron emission tomography (PET) scans: one [18F]FEPPA scan (for translocator protein (TSPO)) and one [11C]SL25.1188 scan (for monoamine oxidase B (MAO-B)) - as well as one magnetic resonance imaging (MRI) scan.

The primary hypotheses are:

1. TSPO total distribution volume (TSPO VT) and MAO-B total distribution volume (MAO-B VT) are greater in the prefrontal cortex (PFC), anterior cingulate cortex (ACC), and hippocampus in COVID-19 with new onset, persistent major depressive episode (MDE) with or without other neuropsychiatric symptoms after recovery from mild respiratory symptoms (DNP-mild).
2. TSPO VT and MAO-B VT are greater in the PFC, ACC, and hippocampus in COVID-19 with new onset, persistent MDE with or without other persistent neuropsychiatric symptoms after recovery from moderate respiratory symptoms (DNP-moderate).

Exploratory hypotheses are:

1. Greater TSPO VT and MAO-B VT in the PFC, ACC, and hippocampus will be positively associated with severity of MDE symptoms and poorer performance on cognitive tasks.
2. TSPO VT and MAO-B VT will be positively correlated in the PFC, ACC and hippocampus in COVID-DNP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Diagnosis of COVID-19
* Recovered from mild or moderate COVID-19 symptoms. Mild is defined as no evidence of pneumonia or hypoxia. Moderate is defined as presence of clinical symptoms of pneumonia but not severe enough to require ongoing use of supplementary oxygen.
* Recovered from physical COVID-19 symptoms including cough, shortness of breath, fever, chills, or gastrointestinal upset for at least 4 weeks
* New onset major depressive episode (MDE) within 3 months after COVID-19, as verified by the Research Version of Structured Clinical Interview for DSM 5 (SCID-5-RV)
* High-affinity-binder (HAB) or mixed-affinity-binder (MAB) genotype for rs6971 polymorphism, based on saliva genetic testing

Exclusion Criteria:

* Lifetime history of an autoimmune disease
* Lifetime history of a neurological disease, excluding migraine
* Lifetime diagnosis of Antisocial or Borderline Personality disorder
* Lifetime history of psychotic symptoms prior to COVID-19
* Lifetime diagnosis of Substance of Alcohol Use Disorder
* Use of street drugs, including marijuana, in the past two months
* Presence of cigarette smoking in the past two months
* Positive urine drug or cotinine screen at any timepoint during the study
* Currently pregnant
* Currently breastfeeding
* Use of aspirin or ibuprofen within the past 2 weeks
* Use of any other anti-inflammatory medication or MAO-B inhibitors within the past 4 weeks
* Use of herbal remedies in the past month
* Presence of metal implant, object or electrical devices that are contraindicated for MRI
* Current disorders of coagulation, blood or ongoing use of anticoagulant medication
* Claustrophobia
* Weight over 400lbs and height over 7ft
* History of undergoing a number of PET scans that will lead participants to exceed the annual (20mSv) / lifetime (8 PET scans) radiation by completing this study
* Current participation in another research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants that have recovered from mild or moderate COVID-19 respiratory symptoms and have a new onset major depressive episode (MDE).
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Translocator protein total distribution volume in prefrontal cortex, anterior cingulate cortex, and hippocampus | within 3 to 4 weeks after initiation of screening
  PET scan measures in DNP-mild and DNP-moderate compared to healthy controls
Monoamine oxidase B total distribution volume in prefrontal cortex, anterior cingulate cortex, and hippocampus | within 3 to 4 weeks after initiation of screening
  PET scan measures in DNP-mild and DNP-moderate compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, M.D., PhD, Principal Investigator — Brain Health Imaging Centre, Centre for Addiction and Mental Health (CAMH)
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No